CLINICAL TRIAL: NCT03359707
Title: Access to Healthcare and the Right to Health of People Living in Disadvantaged Neighborhoods Around Cayenne in French Guiana
Acronym: ACSES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: ACSES
Record Dates: First submitted 2017-11-24; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Health Care Acceptability
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — no intervention just survey

SUMMARY:
ACSES aims to describe the health behaviours and vulnerabilities of poor urban communities living in the greater Cayenne area. It was a questionnaire based study conducted around a red cross truck providing testing.

ELIGIBILITY:
Inclusion Criteria:

* living in poor neighborhoods around cayenne

Exclusion Criteria:

* minors
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: poor populations living in the surroundings of cayenne
Sampling Method: Non-Probability Sample
Enrollment: 696 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Healthcare Acceptability - Questionnaire survey | one year

IPD SHARING:
Plan to Share IPD: No